CLINICAL TRIAL: NCT04449718
Title: Vitamin D Supplementation in Patients With COVID-19: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Vitamin D Supplementation in Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, ROSA MARIA RODRIGUES PEREIRA, Dr, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 30959620.4.0000.0068
Record Dates: First submitted 2020-06-16; First posted 2020-06-29 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
Keywords: COVID-19; vitamin D; acute respiratory syndrome
MeSH Terms: conditions — COVID-19 | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Patients will receive 200,000 IU of vitamin D3 on admission + conventional care
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): Patients will receive an equivalent amount of a placebo solution on admission + conventional care
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — 200,000 IU on admission
  Arms: Experimental
Dietary Supplement: Placebo — 200,000 IU on admission
  Arms: Placebo

SUMMARY:
Coronavirus disease 2019 (COVID-19) was declared an emergency public health problem by the World Health Organization (WHO) in March 2020. Since then, several initiatives by the medical and scientific community have sought alternatives to treat infected individuals, as well as identifying risk or protective factors for the contamination and prognosis of patients. In this perspective, vitamin D supplementation can improve some important outcomes in critically ill patients, being considered a potent immunomodulatory agent. Vitamin D deficiency is a common outcome in critically ill patients, thus making it a modifiable risk factor with great potential for reducing hospital stay and intensive care and mortality. The investigators speculate that vitamin D supplementation could have therapeutic effects in patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of flu syndrome with hospitalization criteria;
* Respiratory rate ≥ 24irpm and / or saturation <93% in room air, or belonging to the risk group for complications: 1. Chronic diseases: heart disease, diabetes mellitus, systemic arterial hypertension and neoplasms, 2. Immunosuppression, 3. Pulmonary tuberculosis; 4. Obesity;
* Tomographic findings compatible with coronavirus disease.

Exclusion Criteria:

* Patient admitted already under invasive mechanical ventilation;
* Patient admitted with severe acute respiratory syndrome and diagnosed with an etiologic agent other than SARS-CoV-2;
* Prior vitamin D supplementation (above 1000 IU/day);
* Renal failure requiring dialysis or creatinine ≥ 2.0mg/dl;
* Admitted patients with expected hospital discharge in less than 24 hours;
* Patient unable to sign the consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
Length of hospitalization | From date of randomization until the date of hospital discharge or death, which is usually less than 1 month
  total number of days that patient remained hospitalized

SECONDARY OUTCOMES:
Mortality | From date of randomization until the date of hospital discharge or death, which is usually less than 1 month
  number of patients that died
Number of cases admitted to Intensive Care Unit (ICU) | From date of randomization until the date of hospital discharge or death, which is usually less than 1 month
  total number of days that patient remained in ICU
Length of use of mechanic ventilator | From date of randomization until the date of hospital discharge or death, which is usually less than 1 month
  total number of days that patient remained in mechanic ventilator
Number and severity of symptoms | From date of randomization until the date of hospital discharge or death, which is usually less than 1 month
Inflammatory markers | Baseline, 14 days after hospitalization and at the moment of hospital discharge or death (usually less than 1 month)
  C-reactive protein, IL-1alpha (pg/ml), IL-1beta (pg/ml), IL-6 (pg/ml), TNF-alpha (pg/ml), IL-1ra (pg/ml), IL-10 (pg/ml) concentration in the serum
C-reactive protein | Baseline, 14 days after hospitalization and at the moment of hospital discharge or death (usually less than 1 month)
  serum concentration
Vitamin D | Baseline, 14 days after hospitalization and at the moment of hospital discharge or death (usually less than 1 month)
  serum concentration
Creatinine | Baseline, 14 days after hospitalization and at the moment of hospital discharge or death (usually less than 1 month)
  serum concentration
Calcium | Baseline, 14 days after hospitalization and at the moment of hospital discharge or death (usually less than 1 month)
  serum concentration
Physical activity | Baseline
  Baecke questionnaire (higher scores mean a higher physical activity level)

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Pereira, PhD, MD, Principal Investigator — School of Medicine, University of Sao Paulo; Bruno Gualano, PhD, Study Director — School of Medicine, University of Sao Paulo
Locations (1):
- Clinical Hospital of the School of Medicine, University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sales LP, Souza LVB, Fernandes AL, Murai IH, Santos MD, Vendramini MBG, Oliveira RM, Figueiredo CP, Caparbo VF, Gualano B, Pereira RMR; in memoriam. Effect of vitamin D3 on antiphospholipid antibodies in hospitalized patients with moderate to severe COVID-19. Clinics (Sao Paulo). 2024 Aug 27;79:100474. doi: 10.1016/j.clinsp.2024.100474. eCollection 2024. PMID 39208655
- [Derived] Fernandes LP, Murai IH, Fernandes AL, Sales LP, Rogero MM, Gualano B, Barroso LP, Milne GL, Pereira RMR, Castro IA. The severity of COVID-19 upon hospital admission is associated with plasma omega-3 fatty acids. Sci Rep. 2024 May 3;14(1):10238. doi: 10.1038/s41598-024-60815-y. PMID 38702342
- [Derived] Fernandes AL, Sales LP, Santos MD, Caparbo VF, Murai IH, Pereira RMR. Persistent or new symptoms 1 year after a single high dose of vitamin D3 in patients with moderate to severe COVID-19. Front Nutr. 2022 Sep 13;9:979667. doi: 10.3389/fnut.2022.979667. eCollection 2022. PMID 36176639
- [Derived] Fernandes AL, Murai IH, Reis BZ, Sales LP, Santos MD, Pinto AJ, Goessler KF, Duran CSC, Silva CBR, Franco AS, Macedo MB, Dalmolin HHH, Baggio J, Balbi GGM, Antonangelo L, Caparbo VF, Gualano B, Pereira RMR. Effect of a single high dose of vitamin D3 on cytokines, chemokines, and growth factor in patients with moderate to severe COVID-19. Am J Clin Nutr. 2022 Mar 4;115(3):790-798. doi: 10.1093/ajcn/nqab426. PMID 35020796
- [Derived] Murai IH, Fernandes AL, Antonangelo L, Gualano B, Pereira RMR. Effect of a Single High-Dose Vitamin D3 on the Length of Hospital Stay of Severely 25-Hydroxyvitamin D-Deficient Patients with COVID-19. Clinics (Sao Paulo). 2021 Nov 26;76:e3549. doi: 10.6061/clinics/2021/e3549. eCollection 2021. PMID 34852148
- [Derived] Stroehlein JK, Wallqvist J, Iannizzi C, Mikolajewska A, Metzendorf MI, Benstoem C, Meybohm P, Becker M, Skoetz N, Stegemann M, Piechotta V. Vitamin D supplementation for the treatment of COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 24;5(5):CD015043. doi: 10.1002/14651858.CD015043. PMID 34029377
- [Derived] Murai IH, Fernandes AL, Sales LP, Pinto AJ, Goessler KF, Duran CSC, Silva CBR, Franco AS, Macedo MB, Dalmolin HHH, Baggio J, Balbi GGM, Reis BZ, Antonangelo L, Caparbo VF, Gualano B, Pereira RMR. Effect of a Single High Dose of Vitamin D3 on Hospital Length of Stay in Patients With Moderate to Severe COVID-19: A Randomized Clinical Trial. JAMA. 2021 Mar 16;325(11):1053-1060. doi: 10.1001/jama.2020.26848. PMID 33595634